CLINICAL TRIAL: NCT02641873
Title: A Phase I Study of BBI608 Administered With FOLFIRI + Bevacizumab in Adult Patients With Metastatic Colorectal Cancer
Brief Title: A Study of BBI608 Administrated With FOLFIRI + Bevacizumab in Adult Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8809001
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic Colorectal Cancer; mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — napabucasin; Fluorouracil; Irinotecan; Leucovorin; Bevacizumab

ARMS (1):
- BBI608 + FOLFIRI +Bevacizumab (Experimental)
  Interventions: Drug: BBI608; Drug: 5-FU; Drug: Irinotecan; Drug: Levofolinate; Drug: Bevacizumab

INTERVENTIONS:
Drug: BBI608 — 240 mg twice daily (480 mg total daily dose)
Drug: 5-FU — 400 mg/m2 bolus will be administered intravenously immediately following irinotecan/levofolinate infusion, followed by 1200 mg/m2/day (total 2400 mg/m2) continuous infusion per cycle(14 days).
Drug: Irinotecan — 180 mg/m2 together with levofolinate will be administered intravenously per cycle(14 days).
Drug: Levofolinate — 200 mg/m2 together with Irinotecan will be administered intravenously per cycle(14 days).
Drug: Bevacizumab — 5 mg/kg will be administered intravenously following irinotecan/levofolinate infusion per cycle(14 days).

SUMMARY:
This is an open-label, multicenter, phase 1 study of BBI608 in combination with FOLFIRI + Bavacizumab. This study population is adult Japanese patients with metastatic colorectal cancers in FOLFIRI + Bevacizumab combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically confirmed advanced unresectable, metastatic or recurrent colorectal carcinoma
2. Evaluable patient by RECISTversion 1.1
3. Stage IV
4. ≥ 20 years of age
5. Life expectancy ≥ 3 months.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
7. Patients with following organ function within 14 days before enrollment (on the basis of the most recent data during the period if multiple data are available)

   * Hemoglobin (Hg) ≥ 9.0 g/dL
   * Neutrophil count ≥ 1.5 x 103/μL
   * Platelet count ≥ 10 x 104/μL
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × institutional upper limit of normal (ULN) [≤ 5 × ULN in presence of liver metastases ]
   * Total bilirubin ≤ 1.5 × institutional ULN [≤ 2 × ULN in presence of liver metastases ]
   * Creatinine ≤ 1.5 × institutional ULN
   * Proteinuria by dipstick urine analysis ≤ 1+. [ UPCR (Urine Albumin-to-Creatinine Ratio) ≤ 1, or protein volume of 24-hour urine collection ≤ 1 g, in the case of patients with a 2+ urine dipstick reading]
8. For female patient of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 30 days after the last protocol treatment dose or 6 months after Bevacizumab treatment.. For male patient of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 90 days after the last protocol treatment dose or 6 months after Bevacizumab treatment
9. Females of childbearing potential have a negative urine pregnancy test
10. Patients who have provided written voluntary consent in person to participate in this study after fully receiving and understanding the information about this study, including study

Exclusion Criteria:

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or hormone therapy, or heart therapy within 21 days of the first dose of BBI608
2. Major surgery within 28 days prior to first dose
3. Have had a brain metastases with a symptom or requiring treatment
4. Have had coinstantaneously active multiple primary cancer
5. Have had a carcinomatous pleural effusion, ascites, or cardiac effusion requiring treatment
6. Crohn's disease, ulcerative colitis, small intestine resection, diarrhea (watery diarrhea), paralysis intestinal, Intestinal obstruction
7. Gastrointestinal perforation, tracheo-oesophageal fistula, fistula
8. Unable or unwilling to swallow BBI608 capsules
9. Uncontrolled inter-current illness (such as Grade 3 active infection, or serious respiratory disease)
10. Uncontrolled hypertension
11. Patients with recent history of hemoptysis of more than 2.5 mL of red blood within 28days before the enrolment
12. Abnormal ECGs which are clinically significant within 28 days before enrolment
13. Patients who are New York Heart Association (NYHA) functional classes III, or IV, or unstable angina
14. Patients newly expressing angina within three months (90 days) before the enrolment
15. Have had myocardial infarction within six months (180 days)before the enrolment
16. Administrating with antiarrhythmic drug
17. Patients who are planning to breast-feeding by whichever 30 days after the last administration of BBI608 or by 6 months after the last administration of Bevacizumab
18. Patients of pregnancy or possibility of pregnancy at current time or possibility of pregnancy within 6 months after the last administration of Bevacizumab
19. Have received other investigational products or not finished the assessment in any clinical study within 28 days before enrollment
20. Known severe hypersensitivity to 5-FU/ levofolinate/ irinotecan/Bevacizumab
21. Administration of atazanavir sulfate
22. Prior treatment with BBI608
23. Ineligible for participation in the study in the opinion of the Investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs) [Safety and Tolerability] | 12 months
  Safety and tolerability assessed by adverse events (AEs), serious adverse events (SAEs)
Number of participants with Dose-limiting toxicities (DLT) [Safety and Tolerability] | 12 months
  Safety and tolerability assessed by determination of unacceptable toxicity in patients.
Cmax (Peak plasma concentration) | Day 1: prior to BBI608 and 2,4,6,8,10,12,24 hours after the first dose.
  Cmax (Peak plasma concentration)
AUC0-24h (Area under the plasma concentration versus time curve) | Day 1: prior to BBI608 and 2,4,6,8,10,12,24 hours after the first dose.
  AUC0-24h (Area under the plasma concentration versus time curve)

SECONDARY OUTCOMES:
Preliminary anti-tumour activity | 6 months(an expected average)
  The radiologic assessments will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST for patients with metastatic colorectal cancer.
Progression Free Survival (PFS) | 12 months
  Participants follow-up for progression free survival will occur. Maximum follow-up time is 12 months after the initial administration of the last subject.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Aichi Cancer Center Hospital, Nagoya, Aichi